CLINICAL TRIAL: NCT04941651
Title: Efficacy of Telenutrition (OBE-COACH) for the Treatment of Overweight Patients With Obesity and/or High Cardiometabolic Risk
Brief Title: Efficacy of Telenutrition for the Treatment of Overweight Patients With Obesity and/or High Cardiometabolic Risk
Acronym: TOOLBAR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: TOOLBAR K160908J
Record Dates: First submitted 2021-06-18; First posted 2021-06-28 (Actual); Last update posted 2024-05-24 (Actual); Status verified 2024-05

CONDITIONS: Overweight and Obesity
Keywords: Overweight patients; Obesity; Cardiometabolic risk; telenutrition; online nutritional coaching service
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- OBE-COACH program (Experimental): The OBE-COACH experimental group: access to the complete OBE-COACH program
  Interventions: Behavioral: OBE-COACH program; Device: Connected devices; Device: Connected Activity Tracer
- e-learning program (Active Comparator): The control group: access to an e-learning program with free access via the web to advice sheets, a menu generator and a catalog of physical activity (resources made available by the site www.mangerbouger.fr ; Public Health France, Ministry of Health) and provision of connected devices (auto-tensiometer and balance).
  Interventions: Device: Connected devices; Device: Connected Activity Tracer; Behavioral: e-learning program

INTERVENTIONS:
Behavioral: OBE-COACH program — OBE-COACH works through private exchanges between the user and an automatic generator of recommendations, advice and messages of encouragement. Web focus groups are propoposed by specialist to respond to the questions of the participants and a tele-interview at 6 months with a dietetician to encourage and assist the patient to make the best use of the program.
  The program is divided into missions to perform. These missions are grouped into 10 families. The completion of each mission and the correct answers to the quiz offer points and bonuses.
  To promote better adherence to the program, missions are not repetitive. They are proposed to surprise the user and constantly renew his desire to connect to the program and achieve goals.
  The intensity level of the program is selected by the user at any time.
  Arms: OBE-COACH program
Device: Connected devices — Connected devices provide to patient are auto-tensiometer and balance. These devices will not be connected to the OBE-COACH program.
  The auto-tensiometer (Tensio-screen, Terraillon) is a connected tensiometer allowing the patient to measure by himself with an armband his systolic and diastolic blood pressure and his heart rate.
  The balance (Web coach premium, Terraillon) is a connected scale to collect body weight.
Device: Connected Activity Tracer — The Activity Tracer (activi-T band, Terraillon) is a a wristband connected activity tracer worn on the wrist that tracks the patient's physical activity and calculates the number of steps, distance traveled and calories burned. The Activity Tracer will not be connected to the OBE-COACH program.
Behavioral: e-learning program — e-learning program with free access via the web to advice sheets, a menu generator and a catalog of physical activity (resources made available by the site www.mangerbouger.fr ; Public Health France, Ministry of Health)
  Arms: e-learning program

SUMMARY:
The OBE-COACH program is an automated online nutritional coaching service that was evaluated in its first version (MXS-CARE program) in a clinical trial coordinated by our team, in type 2 diabetic patients with abdominal obesity. Results have confirmed the efficiency of the program to improve lifestyle habits, including the 4-month diet, and to reduce weight and HbA1c levels.

Based on our experience and the scientific literature, the investigators assume that adherence to the program may diminish in the long term to the point of calling into question its efficiency. So IRIADE compagny developed an enhanced program called OBE-COACH. The OBE-COACH program has been specifically designed to facilitate long-term user adherence. The OBE-COACH program, integrates a bidirectional interactive link between the patient and an automated support system (IRIADE-MED system) associated with an inexpensive remote human support.

In the TOOLBAR study, the investigators will evaluate the efficiency of the OBE-COACH solution in a population of obese patients or overweight persons with at least one cardiometabolic risk factor.

A group of patients will have access to the OBE-COACH program. It will be compared to a control group which will receive an e-learning program with free access to advice sheets via the web, to a menu generator, videos and a catalog of physical activity, (resources made available by the web site www.mangerbouger.fr (public health France, ministry in charge of health) . Indeed, the investigators judged that the loss of patients during follow-up would be greater if e-learning was not offered in the control group.

DETAILED DESCRIPTION:
The management of patients in the TOOLBAR study will be in accordance with French recommendations: a patient who is overweight should benefit from a dietary, physical activity, psychological assistance and medical monitoring advices which can be provided by a general practitioner. In the control group, subjects have access to an e-learning program, including free access via the web to a nutritional information portal and to automated tools providing information and advice for adopting a balanced, low-carb diet and to practice physical activity in line with the guidelines of the national health nutrition plan (PNNS). However, this group will not have access to the OBE-COACH program. The usual follow-up with the attending doctor will be continued.

Patients will be assessed at baseline, 6 months and 12 months. In an ancillary study they could be also assessed at 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Men or women 18 to 75 years
* Obesity defined by a body mass index > 30 kg / m2 or a BMI> 25 kg / m2 with the presence of at least one major cardiometabolic risk factors among the followings: dyslipidemia, hypertension, diabetes, prediabetes
* Stable weight in the last six months (weight variation < 4 kg peak-to-peak)
* Access and current use of internet, possession of an email address and a smartphone.
* Understanding and reading French
* Patient not currently following a nutritional monitoring and not having planned to be engaged in a nutritional monitoring during the coming year

Exclusion Criteria:

* Excessive alcohol consumption > 30 g / day -Pregnant or breastfeeding woman
* symptomatic cardiovascular disease : angina, lower extremity arterial occlusive disease, stroke or myocardial infarction dating of less than 6 months.
* Uncontrolled psychiatric illness
* Patients receiving or about to receive during the study period a systemic or local treatment susceptible to interfere with the evaluation of the primary criteria (corticosteroids, antipsychotics, tricyclic antidepressants) except if these treatments have been stable for at least 6 months without a plan to modify the dose during the 12 months of the study
* Adhering to a prescribed diet for weight loss, in the past 3 months
* Person with a severe eating disorder: bulimia, binge eating disorder according to DSM-V criteria - Presence of celiac disease, Crohn's disease or other metabolic disorder or condition affecting nutritional needs such as allergies or food intolerances (except partial lactose intolerance)
* Anticipated difficulties in following the patient
* Lack of social coverage in France
* Lack of written or electronic informed consent

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 346 (Estimated)
Dates: Start 2024-01-02 (Actual); Primary Completion 2025-11-15 (Estimated); Study Completion 2026-11-15 (Estimated)

PRIMARY OUTCOMES:
Weight reduction of at least 5% between 0 and 12 months. | 12 months
  Weight reduction of at least 5% between 0 and 12 months. The weight, in Kg, will be measured in a state of fastness ≥ 8h, in participants wearing light clothing without shoes on the same scales calibrated at inclusion and 12 months of follow-up.

SECONDARY OUTCOMES:
Weight reduction of at least 5% between 0 and 6 months. | 6 months
  Weight, in Kg, measured in the same conditon at baseline and 6 months.
Weight change between 0 and 6 months | 6 months
  Weight, in Kg, measured in the same conditon at baseline and 6 months.
Weight change between 0 and 12 months | 12 months
  Weight, in Kg, measured in the same conditon at baseline and 12 months.
Waist change between 0 and 6 months | 6 months
  Waist, in cm, measured midway between the last ribs and the anterior superior iliac crest
Waist change between 0 and 12 months | 12 months
  Waist, in cm, measured midway between the last ribs and the anterior superior iliac crest
Triglycerids change between 0 and 12 months | 12 months
  Plasma fasting levels of triglycerides in g/L
HDL cholesterol change between 0 and 12 months | 12 months
  Plasma fasting levels of HDL cholesterol in g/L
LDL cholesterol change between 0 and 12 months | 12 months
  Plasma fasting levels of LDL cholesterol in g/L
non-HDL cholesterol change between 0 and 12 months | 12 months
  Plasma fasting levels of non-HDL cholesterol in g/L (total cholesterol less HDL-C)
Blood glucose change between 0 and 12 months | 12 months
  Plasma fasting levels of glucose in g/L
HbA1c change between 0 and 12 months | 12 months
  Plasma fasting levels of HbA1c in percentage
Systolic blood pressure change between 0 and 12 months | 12 months
  Systolic blood pressure in mmHg as the average of the last 2 automatic measurements out of 3 taken at the level of one arm and spaced about 2 min in the cabinet or by the patient with the auto-tensiometer
Diastolic blood pressure change between 0 and 12 months | 12 months
  Diastolic blood pressure in mmHg as the average of the last 2 automatic measurements out of 3 taken at the level of one arm and spaced about 2 min in the cabinet or by the patient with the auto-tensiometer
Triglycerids change between 0 and 6 months | 6 months
  Plasma fasting levels of triglycerides in g/L
HDL cholesterol change between 0 and 6 months | 6 months
  Plasma fasting levels of HDL cholesterol in g/L
LDL cholesterol change between 0 and 6 months | 6 months
  Plasma fasting levels of LDL cholesterol in g/L
non-HDL cholesterol change between 0 and 6 months | 6 months
  Plasma fasting levels of non-HDL cholesterol in g/L (total cholesterol less HDL-C)
Blood glucose change between 0 and 6 months | 6 months
  Plasma fasting levels of glucose in g/L
HbA1c change between 0 and 6 months | 6 months
  Plasma fasting levels of HbA1c in percentage
Systolic blood pressure change between 0 and 6 months | 6 months
  Systolic blood pressure in mmHg as the average of the last 2 automatic measurements out of 3 taken at the level of one arm and spaced about 2 min in the cabinet or by the patient with the auto-tensiometer
Diastolic blood pressure change between 0 and 6 months | 6 months
  Diastolic blood pressure in mmHg as the average of the last 2 automatic measurements out of 3 taken at the level of one arm and spaced about 2 min in the cabinet or by the patient with the auto-tensiometer
Change in adherence to the Mediterranean diet : Score PREDIMED | 12 months
  Change between 0 and 12 months of adherence to mediterranean diet,evaluated by the dietetic score PREDIMED (validated checklist of 14 items). Higher scores indicate greater adherence to the diet assigned
Change in adherence to the Mediterranean diet : fruits and vegetables consumption | 12 months
  Change between 0 and 12 months in terms of perrcentage of consumption of fruits and vegetables on the recommended 400 g/day
Change in adherence to the Mediterranean diet : Score PREDIMED | 6 months
  Change between 0 and 6 months of adherence to mediterranean diet,evaluated by the dietetic score PREDIMED (validated checklist of 14 items). Higher scores indicate greater adherence to the diet assigned
Change in adherence to the Mediterranean diet : fruits and vegetables consumption | 6 months
  Change between 0 and 6 months in terms of percentage of consumption of fruits and vegetables on the recommended 400 g/day
Change between 0 and 12 months of Energy intake | 12 months
  Energy intake, in Kcal/day, evaluated with the validated NAQA questionnaire
Change between 0 and 12 months of proteins intake, in g/day, evaluated with the validated NAQA questionnaire | 12 months
Change between 0 and 12 months of sucrose intake in g/day, evaluated with the validated NAQA questionnaire | 12 months
Change between 0 and 12 months of lipids intake in g/day, evaluated with the validated NAQA questionnaire | 12 months
Change between 0 and 12 months of cholesterol intake | 12 months
  Cholesterol intake, in mg/day, evaluated with the validated NAQA questionnaire
Change between 0 and 12 months of calcium intake in mg/day, evaluated with the validated NAQA questionnaire | 12 months
Change between 0 and 12 months of sugary drinks consumption in number of glasses/day | 12 months
Change between 0 and 12 months of alcohol drinks consumption in number of glasses/day | 12 months
Change between 0 and 6 months of sugary drinks consumption in number of glasses/day | 6 months
Change between 0 and 6 months of alcohol drinks consumption in number of glasses/day | 6 months
Change between 0 and 12 months of tobacco consumption in number of cigarettes/day | 12 months
Change between 0 and 6 months of tobacco consumption in number of cigarettes/day | 6 months
Change between 0 and 12 months of Adherence to the WHO recommendations for physical activity, measured in Metabolic Equivalent of Task, MET, evaluated with the GPAQ questionnaire. | 12 months
Change between 0 and 6 months of Adherence to the WHO recommendations for physical activity, measured in Metabolic Equivalent of Task, MET, evaluated with the GPAQ questionnaire. | 6 months
Adherence to OBE-COACH program at 12 months, evaluated by the average percentage of questions (sent by IRIADE) with replies from the subject per week during the previous month. | 12 months
Adherence to OBE-COACH program at 12 months, evaluated by the number of participation in web focus groups over the last 6 months. | 12 months
Adherence to OBE-COACH program at 6 months, evaluated by the average percentage of questions (sent by IRIADE) with replies from the subject per week during the previous month. | 6 months
Adherence to OBE-COACH program at 6 months, evaluated by the number of participation in web focus groups over the last 6 months. | 6 months
Change between 0 and 12 months of Food impulsivity evaluated by the TFEQ21 questionnaire | 12 months
Change between 0 and 6 months of Food impulsivity evaluated by the TFEQ21 questionnaire | 6 months
Evolution between 0 and 12 months of Symptoms of anxiety, measured with the HAD questionnaire (score 0 to 21) | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Marylou Para, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital La Pitié Salpêtrière, Paris, France

IPD SHARING:
Plan to Share IPD: Yes
Data are available upon reasonable request. The procedures carried out with the French data privacy authority (CNIL, Commission nationale de l'informatique et des libertés) do not provide for the transmission of the database, nor do the information and consent documents signed by the patients.
  Consultation by the editorial board or interested researchers of individual participant data that underlie the results reported in the article after deidentification may nevertheless be considered, subject to prior determination of the terms and conditions of such consultation and in respect for compliance with the applicable regulations.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning 3 months and ending 3 years following article publication. Requests out of these time frame can also be submitted to the sponsor
Access Criteria: Researchers who provide a methodologically sound proposal